CLINICAL TRIAL: NCT05689996
Title: Effect of Using of Ozone-based Eye Drops as Adjuvant Therapy in the Management of Microbial Keratitis in Comparison to the Conventional Therapy
Brief Title: Ozone-based Eye Drops as Adjuvant Therapy in Microbial Keratitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abeer Abdel-Fattah Mohammed Ali, Ophthalmology Resident, Assiut University Hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ozone-based eye drops
Record Dates: First submitted 2021-10-11; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Keratitis
Keywords: Microbial keratitis
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Intervention Model Description: Preparation of nanostructure lipid carriers (NLCs):
  The emulsification-solvent evaporation technique was used to prepare the NLCs. The method was followed by ultrasonication as reported [1]. In brief, the lipid phase was composed of stearic acid (solid lipid, 300 mg and oleic acid (liquid lipid, 300 mg) dissolved in ethanol (2 mL, 1:1, v/v) at 70oC. In total, 20 mL of the distilled water containing 2% of the Tween® 80 were heated at 70 oC to prepare the aqueous phase. Then, both phases, aqueous and lipid phases, were mixed at the same temperature using 2000 rpm stirring for 15 min. The resulting pre-emulsion obtained from the mixture of the aqueous and lipid phases was sonicated by a probe-type sonicator (Cole-Parmer, Vernon Hills, IL, USA) for 10 min at pulse-ON for 3 s and pulse-OFF for 5 s (40 W). The obtained dispersion was allowed to cool to RT under continuous stirring for 60 min at 1000 rpm for 1 h to obtain the NLCs dispersions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infective keratitis (Experimental): Preparation of nanostructure lipid carriers (NLCs):
  The emulsification-solvent evaporation technique was used to prepare the NLCs. The method was followed by ultrasonication as reported [1]. In brief, the lipid phase was composed of stearic acid (solid lipid, 300 mg and oleic acid (liquid lipid, 300 mg) dissolved in ethanol (2 mL, 1:1, v/v) at 70oC. In total, 20 mL of the distilled water containing 2% of the Tween® 80 were heated at 70 oC to prepare the aqueous phase. Then, both phases, aqueous and lipid phases, were mixed at the same temperature using 2000 rpm stirring for 15 min. The resulting pre-emulsion obtained from the mixture of the aqueous and lipid phases was sonicated by a probe-type sonicator (Cole-Parmer, Vernon Hills, IL, USA) for 10 min at pulse-ON for 3 s and pulse-OFF for 5 s (40 W). The obtained dispersion was allowed to cool to RT under continuous stirring for 60 min at 1000 rpm for 1 h to obtain the NLCs dispersions.
  Interventions: Drug: Ozone-Based Agent

INTERVENTIONS:
Drug: Ozone-Based Agent — Ozone-based eye drops as adjuvant therapy in microbial keratitis
  Other Names: ozone-based eye drops

SUMMARY:
To compare the therapeutic effect of ozone-based eye drops as an adjuvant therapy to that of the conventional topical antimicrobial agents in patients with microbial keratitis . The therapeutic response will be evaluated with clinical examination follow up .

DETAILED DESCRIPTION:
Inflammatory corneal diseases remain a major challenge in ophthalmology , for example microbial keratitis still remains a serious cause of corneal opacity and subsequently visual impairment worldwide [1,2,3 ]. Rarely the infection occurs in the normal eye as the human cornea has its natural resistance against infection. However, predisposing factors such as pre-existing corneal disease, contact lens wear , aggressive topical antimicrobial therapy , prior ocular surgery , ocular surface disease, and trauma may change the defense mechanisms of the ocular surfaces and thereafter permit entry of different pathogens. Treatment aims to managing any other associated ocular surface disease involvement, removing any known risk factors in addition to antimicrobial therapy . The patient requires close treatment response monitoring, sometimes including hospitalization followed by frequent outpatient visits. The risk of developing microbial keratitis and the severity of the disease depend on both the type of the infecting organism and the condition of the ocular surface .[4] .It is important to confirm infection in order to determine the most effective treatment, especially at the initial stage when the treatment is not based on culture results. Microbial keratitis is treated by topical eye drops containing anti-inflammatory and anti- bacterial agents. The current antimicrobial treatments often lack efficacy because infections occur in hypoxic tissue contain methicillin-resistant Staphylococcus aureus and Pseudomonas aeruginosa so new products for the treatment of ocular inflammation and pain are needed. In addition, Increased bacterial antibiotic resistance contributes to the use of a therapy based on natural products, such as ozonized oil, which have a wide spectrum of antimicrobial effects for therapeutic applications.

The use of ozone in anterior segment pathologies could be providential due to its anti-inflammatory and bactericidal activity by direct oxidation mediated by lipoperoxyde and hydrogen peroxide, selective cytotoxicity on fast dividing cells, through bacterial lysis then cell death and negative regulation on mitochondrial activity in bacteria.[5] .Ozone dose trigger several useful biochemical mechanisms and reactivate the antioxidant system (i.e., catalase, superoxide dismutase, glutathione peroxidase, etc.) [ 6] in addition to promoting tissue repair properties , assumed to be due to the upregulation of platelet-derived growth factor, transforming growth factor-β, and vascular endothelial growth factor expressions. Eye drops containing ozone were recently used in the management of ocular surface infection caused by bacteria, viruses and fungi, [ 7-9] and a specific formulation containing liposomal ozonated sunflower oil (Ozodrop®, FB Vision, San Benedetto del Tronto, Italy) that is well tolerated by the ocular surface has been developed. [ 10 ] Ozone in the gaseous state is extremely reactive and not always suitable as a topical treatment. In saline solution, its concentration reduces quickly with a first-order kinetics and its half-life is 2 h: this means that in about 24 h very little ozone will be remains in the solution . In spite of its instability, the ozone molecule can be stabilized - for topical use - as an ozonide, an organic analog of ozone, formed by the reaction of ozone with an unsaturated fatty acid , such as oleic acid [ 12-11] . The zone eye drops will be used at regimen of 3 times per day in addition of antibiotics eye drops.

To superintend its effectiveness in dealing with microbial keratitis , assessment of visual acuity outcome , clinical examination , a follow up imaging from slit lamp will be done and an imaging modality as Anterior segment optical coherence tomography (ASOCT ) can be done . ASOCT is a relatively new imaging modality in the imaging field towards a better evaluation, diagnosis and management of many anterior segment diseases [13,14] .Current uses of ASOCT are corneal thickness evaluation , depth of corneal deposits and lesions including dystrophies, details of corneal inflammation, dry eye evaluation and diagnosis of surface neoplasia in early stages [ 15].Its purpose in this study is to describe the ASOCT cornea features during active stage of microbial keratitis and to evaluate its contribution for its diagnosis and the follow-up Images acquired by AS OCT will be compared to the clinical assessment .

ELIGIBILITY:
Inclusion Criteria:

* Patients with active microbial keratitis ( bacterial , viral or fungal )
* with positive culture and sensitivity result
* Any age group.
* accepting well informed consent for using the ozone eye drops

Exclusion Criteria:

* patients refuse to participate
* Patients with other forms of keratitis rather than infective keratitis . patients who will not complete treatment .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Ozone-based eye drops as adjuvant therapy in microbial keratitis | at 48 hours , 2-3 weeks
  compare the therapeutic effect of ozone-based eye drops as an adjuvant therapy to that of the conventional topical antimicrobial agents in patients with microbial keratitis.
  Main outcome measurements include decrease in size, depth and infiltrate of the ulcer in millimeters measured on slit lamp biomicroscopy .

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spadea L, Tonti E, Spaterna A, Marchegiani A. Use of Ozone-Based Eye Drops: A Series of Cases in Veterinary and Human Spontaneous Ocular Pathologies. Case Rep Ophthalmol. 2018 May 24;9(2):287-298. doi: 10.1159/000488846. eCollection 2018 May-Aug. PMID 29928225
- [Background] Paduch R, Urbanik-Sypniewska T, Kutkowska J, Choragiewicz T, Matysik-Wozniak A, Zweifel S, Czarnek-Chudzik A, Zaluska W, Rejdak R, Toro MD. Ozone-Based Eye Drops Activity on Ocular Epithelial Cells and Potential Pathogens Infecting the Front of the Eye. Antioxidants (Basel). 2021 Jun 16;10(6):968. doi: 10.3390/antiox10060968. PMID 34208703
- [Background] Passidomo F, Pignatelli F, Addabbo G, Costagliola C. Topical Liposomal Ozonated Oil in Complicated Corneal Disease: A Report on Three Clinical Cases. Int Med Case Rep J. 2021 May 14;14:327-332. doi: 10.2147/IMCRJ.S311839. eCollection 2021. PMID 34017203
- [Background] Sridhar MS, Martin R. Anterior segment optical coherence tomography for evaluation of cornea and ocular surface. Indian J Ophthalmol. 2018 Mar;66(3):367-372. doi: 10.4103/ijo.IJO_823_17. PMID 29480245